CLINICAL TRIAL: NCT03986658
Title: Dose-Response Study of Linear Asymmetric rTMS in Adolescent Treatment-Resistant Depression: Tolerability of Treatment Durations Ranging From Ten Days to One Day
Brief Title: Linear Asymmetric rTMS in Adolescent Treatment-Resistant Depression: Tolerability of Treatment Durations Ranging From Ten Days to One Day
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NeuroQore Inc. (Industry)
Collaborators: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEO19P1
Record Dates: First submitted 2019-05-31; First posted 2019-06-14 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Treatment Resistant Depression
Keywords: Major Depressive Disorder; Repetitive Transcranial Magnetic Stimulation (rTMS); Treatment-Resistant Depression; Adolescents
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: rTMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents (Experimental): Device: First Dawn rTMS System used in 18 patients divided into groups of 3. Each group will receive a different and gradually increasing frequency of treatment sessions/day (1-10) over a decreasing number of days (10-1). The total number of pulses for all levels will be 30,000. The use of each level will be dependent on tolerability and safety of the previous lower level, i.e., if one level is not tolerated well by a group, progression to the next level will not occur.
  Interventions: Device: Linear Asymmetric rTMS System

INTERVENTIONS:
Device: Linear Asymmetric rTMS System — Linear Asymmetric rTMS System

SUMMARY:
This is a pilot interventional study to investigate the acceptability, tolerability, and side effect profile for varying numbers of treatment sessions/day of a new rTMS treatment in adolescents with treatment-resistant depression (TRD). Conventional rTMS has been limited to sinusoidal biphasic electromagnetic pulses. In contrast, the First Dawn rTMS system by NeuroQore can sustain a repetitive linear asymmetric pulse. In addition, identification of rTMS treatment sites in adolescents with TRD most often relies on anatomic landmarks, but the First Dawn rTMS system utilizes personal fMRI data in a novel algorithm to determine where to apply the rTMS in each patient.

Based on adult data in healthy volunteers and patients with TRD, the investigators propose that the First Dawn rTMS system will be acceptable and well-tolerated by adolescents and will have minimal side effects. Please see https://clinicaltrials.gov/ct2/show/NCT02667041 for details on the completed pilot study in adults.

The investigators aim to investigate acceptability, tolerability, and side effects in groups of patients receiving treatment in numbers of sessions/day that are gradually accelerated over the course of the study. Results will be used to inform the development of a randomized controlled trial.

DETAILED DESCRIPTION:
The 18 patients will be placed into 6 sub-groups sequentially as they are enrolled. All patients will receive a maximum of 30,000 pulses in their treatment course, as tolerated. The first group will receive daily sessions, similar to standard rTMS treatment. Each of the remaining groups will be set to receive more frequent sessions/day in decreasing numbers of days on a graduated schedule while holding the total number of pulses for each patient's treatment course at 30,000 pulses. in addition, the investigators will recruit one healthy volunteer to test fMRI server data transfer and analysis. This healthy volunteer will not receive rTMS.

Primary Objectives

The primary objectives of this study are to assess: 1) the feasibility of enrollment (number of patients who enroll divided by the number of patients approached), 2) study retention (number of patients completing the study divided by the number enrolled), and 3) AE/SE profile of the treatment at each protocol level and 4) patient experience in the study across the sample and within the sub-groups.

Secondary Objectives

The secondary objectives of this study are to: 1) evaluate daily changes in symptoms of depression and mental status; 2) evaluate fMRI changes in the LDLPFC after treatment; 3) evaluate post-treatment and 3-month changes in depression symptoms, global function, mental status, verbal memory.

ELIGIBILITY:
Inclusion:

1. Meets criteria for DSM-5 MDD, as determined by a structured psychiatric interview.
2. Meets criteria for TRD:

   1. failed two adequate courses of antidepressant medication OR
   2. failed adequate course of medication AND one course of psychotherapy.
3. Score of > 40 on Child Depression Rating Scale-Revised OR score of > 20 on Child Depression Inventory-2.
4. Fluent in speaking and reading English.

Exclusion:

1. Positive pregnancy test.
2. Current or past: bipolar disorder, psychotic disorder, autism spectrum disorder, intellectual disability, substance use disorder, conduct disorder, as determined by a structured psychiatric interview.
3. Medical illness that could lower the seizure threshold, e.g., epilepsy from any cause.
4. Medications that could lower the seizure threshold or affect brain function.
5. Psychotropic medications changed in two weeks prior to enrollment.
6. Fails the TMS safety screening questionnaire.
7. Fails fMRI screening process.
8. Left-handed (may indicate different cortical lateralization which could affect outcomes).
9. Involuntarily committed to the hospital.

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient Enrollment Rate | Through study completion, an average of 10 months
  Number of patients who give consent divided by the number who are approached.
Patient Completion Rate | Through study completion, an average of 10 months
  Number of patients who complete the study divided by the number of patients who enroll in the study.
Side Effects Profile | Through study completion, an average of 10 months
  Measured with the rTMS Side Effect Questionnaire
Patient Experience | Through study completion, an average of 10 months
  Measured with the Multi-Care Institute for Research and Innovation Research Participant Satisfaction Questionnaire

SECONDARY OUTCOMES:
Change in self-reported MDD symptoms | Change from baseline score to score at 3 months
  Measured with the Child Depression Inventory-2.(CDI-2)
Change in clinician-rated MDD symptoms | Change from baseline score to score at 3 months
  Measured with the Child Depression Rating Scale-Revised (CDRS-R)
Change in function | Change from baseline score to score at 3 months
  Measured with the Children's Global Assessment Scale (C-GAS)
Change in mental status | Change from baseline score to score at 3 months
  Measured with the Mini-Mental State Examination (MMSE)
Change in short-term verbal memory | Change from baseline score to score at 3 months
  Measured with the Hopkins Verbal Learning Test-Revised (HLVT-R)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Pajer, MD, Principal Investigator — Children's Hospital of Eastern Ontario (CHEO)
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
clintrials.gov